CLINICAL TRIAL: NCT05045690
Title: BREATHE: An Efficacy-implementation Trial of a Brief Shared Decision Making Intervention Among Black Adults With Uncontrolled Asthma in Federally Qualified Health Centers (Pre-Trial)
Brief Title: BREATHE: An Efficacy-implementation With Listening Sessions
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Clinical Directors Network (Network); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Maureen George, Professor of Nursing at the Columbia University Medical Center, Columbia University
Other Study IDs: AAAT0939 - pre-trial; 1R01NR019275 (NIH)
Record Dates: First submitted 2021-09-07; First posted 2021-09-16 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Listening sessions: The research team will collect qualitative data from the listening sessions (focus groups) using a semi-structured iterative focus group guide.

DETAILED DESCRIPTION:
The trial will be informed by 4-8 listening sessions (research focus groups) with 4-8 adults with asthma at each of four sites (N=32). The trial will also include interviews with approximately 1-2 providers and 1-2 administrators at each site (N=8-16).

Adults with asthma and providers/administrators will participate in pre-trial listening sessions (focus groups) prior to recruiting for other phases in this project. They will share their experience with asthma and clinical research. This will aid in gaining the identification of possible barriers to participation and will provide the opportunity for the patients and providers/administrators to identify which of the planned outcomes they consider to be most meaningful. After obtaining informed consent from participants, the research team will collect demographic and diagnosis information, administer surveys and conduct listening sessions.

The research team will collect demographic information and administer questionnaires to characterize the participants. These include: Demographic form, Asthma history (patient), Asthma history (family), Asthma Control Questionnaire, Shared Decision Making Questionnaire, Medication Adherence Record Scale (preventer), Conventional and Alternative Management for Asthma (patient), Conventional and Alternative Management for Asthma (family), Asthma Quality of Life Questionnaire, Newest Vital Sign, and Short Assessment of Health Literacy. Pre-trial listening sessions: one 2-hour session.

Providers/administrators will participate in one 30-minute session interview.

This pre-trial is an informative research that will help design an RCT with masking and allocation in the future.

ELIGIBILITY:
Inclusion Criteria:

1. be adults (> 18 years of age or emancipated)
2. self-report 'black' race (African American, African, Caribbean, West Indian, multi-racial [black AND one or more additional races]); identify their ethnicity as Hispanic OR non-Hispanic
3. have clinician-diagnosed asthma
4. receive asthma care at a partner federally-qualified health center (FQHC)

Exclusion Criteria:

1. non-English speaking
2. serious mental health conditions that preclude completion of study procedures or confound analyses
3. participation in a listening session

Inclusion Criteria (provider/administrator): Providers who manage a panel of adult asthma patients (i.e., eligible for randomization in the trial) and administrators at that site will be recruited to participate in the interviews.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from federally qualified health centers (FQHCs)
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-11-19 (Actual); Primary Completion 2022-06-09 (Actual); Study Completion 2022-06-09 (Actual)

PRIMARY OUTCOMES:
Number of participants who completed listening sessions | Visit 1 (approximately 120 minutes)
  Listening sessions (research focus groups) will be held pre-trial to explore experiences with asthma and clinical research. Sharing from these sessions will be observational in nature where information will be collected to aid the design/implementation of other portions in this project.
Number of participants who completed clinician/administrator pre-trial interviews | Visit 1 (approximately 30 minutes)
  Interviews will be held pre-trial to explore experiences with asthma and clinical research. Sharing from these sessions will be observational in nature where information will be collected to aid the design/implementation of other portions in this project.

CONTACTS AND LOCATIONS:
Overall Officials: Maureen T George, PhD, Principal Investigator — Columbia University
Locations (1):
- Clinical Directors Network, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided